CLINICAL TRIAL: NCT06873139
Title: FIT4Life Text Message Program
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Jordan Carlson, Director, Community-Engaged Health Research, Principal Investigator, Children's Mercy Hospital Kansas City
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STUDY00003517
Record Dates: First submitted 2025-02-20; First posted 2025-03-12 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Physical Activity; Behavior Change
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High Arm (Experimental): High-arm participants will receive daily messages related to wear reminders, encouragements, congratulatory content, and behavior change based on the activity tracker data. Step counts from the activity tracker are included in some messages to track and facilitate step goals. Some text message content asks for a response from the participant to help tailor later messages for behavior change support.
  Interventions: Behavioral: text messages
- Low Arm (Experimental): Low arm participants will receive weekly messages related to reminders to wear their activity tracker and tips on how to use the tracker.
  Interventions: Behavioral: text messages

INTERVENTIONS:
Behavioral: text messages — There will be two arms for the texting intervention: high and low. Both arms will receive text messages, but the frequency of the messages will vary by arm. Text intervention messaging will be sent through an automated text messaging service programmed by the CM Research Informatics team, which has been approved by the institution.

SUMMARY:
FIT4Life is a text message based physical activity project that includes one baseline week and 26 weeks of intervention delivery. Study participants will be provided with fitness trackers to support their physical activity goals. The text messages are intended to motivate participants to engage in physical activity throughout the week, but do not prescribe specific exercises/workout regimens for participants to follow.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Able to read, write, and speak English
* Currently a Diabetes Prevention Program group or in a similar group that is recruited by the external community partner (Our Healthy Jackson County)

Exclusion Criteria:

* Does not meet the inclusion criteria listed above

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Acceptability and preferences | From enrollment to the end of program at 27 weeks
  Descriptive analyses will be used to analyze the survey data and qualitative thematic analyses will be used to analyze interview data to determine participant preferences and program acceptability.

SECONDARY OUTCOMES:
Change in Physical Activity Minutes | From enrollment to the end of program at 27 weeks
  Longitudinal models will be used to investigate changes in physical activity minutes over time, from before (baseline) to after the intervention.
Change in Physical Steps | From enrollment to the end of program at 27 weeks
  Longitudinal models will be used to investigate changes in steps over time, from before (baseline) to after the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Kansas City Community, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
Participant data will be aggregated and shared to protect privacy.